CLINICAL TRIAL: NCT05784350
Title: Preoperative Point of Care Ultrasound Guided Fluid Optimization and Intravenous Ondansetron to Prevent General Anesthesia-Induced Hypotension: A Randomized Controlled Trial
Brief Title: Preoperative Point of Care Ultrasound Guided Fluid Optimization and Intravenous Ondansetron to Prevent General Anesthesia-Induced Hypotension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0068-23-MMC
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Intra-operative Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous fluid bolus (Active Comparator)
  Interventions: Drug: fluid boluses guided by IVC diameter via US/administration of pre-operative IV Odansetrone
- Intravenous Ondansetron (Active Comparator)
  Interventions: Drug: fluid boluses guided by IVC diameter via US/administration of pre-operative IV Odansetrone
- No intervention (No Intervention)

INTERVENTIONS:
Drug: fluid boluses guided by IVC diameter via US/administration of pre-operative IV Odansetrone — group A will undergo fluid repletion guided by their IVC-CI - if a collapsible IVC, defined as a CI equal or greater than 43%, is observed, patients will receive repeated Lactated Ringer's 500 ml boluses followed by repeated IVC-CI measurements until their CI is less than 43%, and up to 1.5L.
  Group B will undergo the same intervention, with the addition of intravenous ondansetron 4 mg in 10 ml normal saline 20 minutes before induction of general anesthesia.
  Arms: Intravenous Ondansetron; Intravenous fluid bolus

SUMMARY:
Hypotension is a common side-effect of general anesthesia induction and is related to adverse outcomes including significantly increasing risk of one-year mortality. Even short durations of intraoperative hypotension have been associated with acute kidney injury (AKI) and myocardial injury.Half of all the patients were fluid-responsive, pointing to volume status as a significant risk factor. Ultrasound measurements of inferior vena cava (IVC) diameter with respiration, including the maximal diameter of the IVC (dIVCmax) at the end of expiration during spontaneous respiration and the collapsibility index (CI), have been recommended as rapid and noninvasive methods for estimating volume status.

In attempt to prevent hypotension after spinal anesthesia induction, Ondansetron, a serotonin receptor antagonist, has been used effectively .

Research Question Can preoperative IVC-US guided fluid optimization and intravenous ondansetron reduce the incidence of general anesthesia-induced hypotension in adult patients undergoing elective non-cardiac non-obstetric surgery?

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Elective, non-cardiac, non-obstetric surgery under general anesthesia
3. American Society of Anesthesiologists physical status classification I - III

Exclusion Criteria:

1. MAP below 60 mmhg prior to the induction of general anesthesia.
2. Patients treated with angiotensin converting enzyme inhibitors (ACE-I) or angiotensin receptor blockers (ARB) on the day of surgery.
3. Patients with heart failure with ejection fraction (EF) < 40%.
4. Patients with documented acute or chronic renal failure.
5. Patients with hepatic failure.
6. Patients with neuraxial (spinal/epidural) anesthesia performed before induction of general anesthesia.
7. Patients with suspected difficult airway.
8. Patients with documented allergy to Ondansetron or prolonged QT-syndrome.

   -

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of preoperative IVC-guided fluid optimization and intravenous ondansetron in reducing the incidence of hypotension after the induction of general anesthesia | 5 years
  To determine the efficacy of preoperative IVC-guided fluid optimization and intravenous ondansetron in reducing the incidence of hypotension after the induction of general anesthesia in adults presenting for elective non-cardiac, non-obstetric surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No